CLINICAL TRIAL: NCT03586895
Title: e-Connect: A Service System Intervention for Justice Youth at Risk for Suicide
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: George Mason University (Other); National Institute of Mental Health (NIMH) (NIH); Chestnut Health Systems (Other)
Responsible Party: Principal Investigator, Katherine Elkington, Professor of Clinical Medical Psychology (in Psychiatry), Columbia University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AAAU8900; R01MH113599 (NIH)
Record Dates: First submitted 2018-06-21; First posted 2018-07-16 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Suicide
Keywords: Suicidal Behavior; Behavioral Health Problems; e-Connect
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: pre-post design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-Connect (Experimental): County receives training and materials and subsequently begins the e-Connect intervention
  Interventions: Behavioral: e-Connect
- Standard of care (No Intervention): Counties use the standard of care and there is no intervention in practices.

INTERVENTIONS:
Behavioral: e-Connect — e-Connect
  Arms: e-Connect

SUMMARY:
The investigators propose to create e-Connect, a new service delivery model that will enable real time identification and targeted, county-specific referral and linkage of participants with suicidal behavior (SB) and related behavioral health (BH) problems. e-Connect will: (i) establish and formalize interagency referral decisions based on clinical need, jointly derived by JJ (juvenile justice) and BH agencies; (ii) train probation staff to increase BH/SB understanding; (iii) utilize an existing evidence-based (EB) BH/SB screen; and (iv) develop a mobile application to seamlessly integrate screening, classification of clinical need and development of a related referral plan. There are 4 project phases: Development, Baseline, Implementation, and Sustainment/Evaluation. After development, activities take place in 10 NY (New York) counties and all study counties will begin the intervention at the same time. The investigators will examine changes in outcomes (e.g., service use) relative to baseline in (i) identification of participants service need (SB and BH correlates) in juvenile probationers; (ii) cross-system (probation-BH agency) referral; and (iii) participants BH service use (access and engagement). Analyses will further consider contributions of multi-level factors (e.g., staff, organizational, family, and community) that influence implementation (feasibility, acceptability, sustainability) of e-Connect across various probation department processing categories (e.g. status offenders, diversion cases). The investigators will consider the role of mediating elements (e.g., probation practices) in explaining the association between e-Connect and identification, referral, and service use.

DETAILED DESCRIPTION:
While youth at all juvenile justice (JJ) processing points are at increased risk for suicidal behavior (SB) and associated behavioral health (BH) issues, those supervised in community settings (e.g., probation), may be at greatest risk: (a) protocols for identification and service referral are far more common in secure settings, (b) national policy increasingly favors community supervision/diversion over incarceration, (c) participants supervised in the community have far more access to means and opportunity than do those in secure settings, and (d) the multi- system coordination challenges to accessing BH care for community JJ participants are far greater than for those secure care. The investigators propose to adapt and test the utility of a multi-level service delivery model that increases identification of SB and related BH problems, guides targeted referral, trains staff and structures interagency collaboration to increase uptake of BH services by participants on probation; and document the organizational elements required to widely-implement this model in juvenile probation and community treatment settings. The model is based on our earlier, evidence-based linkage protocols from Project Connect, and capitalizes on technological advances unavailable at Connect's 2007 development, so as to address earlier implementation issues. Working in 10 NYS counties, project specific aims are (1) to develop technologically advanced cross-system identification/linkage service model that trains staff, formalizes interagency collaboration and referral decision-making and uses a mobile application to seamlessly combine (a) screening for SB and related BH problems, (b) classification of clinical need and (c) county-specific streamlined referral plans for BH services; (2) to examine the degree to which, compared to Baseline, e- Connect improves (a) intermediary PO practice outcomes (service need identification, cross-system referral) and increasing (b) participants BH service use (access, engagement); and (3) to elucidate multi-level factors (e.g., staff, organizational, participants/family, community,) that influence implementation (feasibility, acceptability, sustainability) of e-Connect across various probation department processing categories (e.g. status offenders, diversion cases) to inform comprehensive scale-up. The theoretically based mechanisms (e.g., changes in staff knowledge and self-efficacy; agency structural characteristics) by which PO practice change affects BH service use will also be examined. Guided by the GPM and CFIR framework, this 5-year study will comprise 4 project phases: (1) Development, (2) Baseline data collection, (3) Implementation, and (4) Sustainment. After development, it was originally planned that counties would be randomized to one of 4 Waves to begin implementation of e-Connect at 4-month intervals in a stepped-wedge design. Implementation activities continue for 18m and sites' use of e-Connect protocols after 18m will be an indication of sustainability. However, at the beginning of the trial, the state in which the current study was implemented introduced the raise the age policy requiring all adjusted youths on probation to receive an evidence-based BH screen. Thus, in order to be compliant with state mandates, all study counties had to begin the intervention at the same time, requiring a 'flattening' of the step-wedge design into a simple pre-post design. Due to this change, analyses were simplified as described in the statistical analysis section. This initiative is one of the first to address SB and advance JJ participants enrollment in BH treatment. Because the investigators propose addressing risk and acute SB, this study has the likelihood of identifying and linking to services high-risk, high need participants that are often overlooked.

ELIGIBILITY:
Sample: County Probation Leadership (Executive and Supervisory) and Line (Juvenile Probation Officers) Staff

Inclusion Criteria: Probation Officers ages 21-70 years old with active employment at the probation department working with youth, or supervise those working with youth in one of the following capacities: probation supervision, assessment, and referral, or engage in work that is related to policies, procedures, and decisions around these activities in 10 site counties

Exclusion Criteria: There are no exclusionary criteria and no special classes of participants.

Sample: Youth on Probation

Inclusion Criteria: All new intakes ages 10-18 years old

Exclusion Criteria: There are no exclusionary criteria and no special classes of participants.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12838 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral health treatment initiation | Monthly in years 2- 5
  Date of first behavioral health appointment/contact extracted from state management information system (MIS)

SECONDARY OUTCOMES:
Behavioral health referral | Day one of probation
  Clinically appropriate referral made by probation officer to behavioral health provider, based on screening results, indicated by referral date extracted from MIS
Youth screened for risk of suicide | Day one of probation
  Evidence-based screening tool self administered by youth
Family Experience and Fidelity of e-Connect | Bimonthly years 2-5
  PO completes family debriefing checklist: family receptivity to screening results and referral plan
e-Connect Sustainability | end of implementation through sustainment period, monthly
  Ongoing use of e-Connect during post implementation phase

OTHER OUTCOMES:
Suicidal Behavior, Non-Suicidal Self-Injury (NSSI), BH knowledge | Years 1-5
  Measured during pre-post quizzes following web-based training modules; developed for study
Perceived importance of screening and referral to BH - Baseline Phase services | 2 months
  Subscales for screening - Measure assessing perceived importance of activities associated with screening, referral and linkage - developed by JJTRIALS research cooperative.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Elkington, PhD, Principal Investigator — Columbia University/New York State Psychiatric Institute
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wasserman GA, Elkington KS, Robson G, Taxman F. Bridging juvenile justice and behavioral health systems: development of a clinical pathways approach to connect youth at risk for suicidal behavior to care. Health Justice. 2021 Nov 29;9(1):36. doi: 10.1186/s40352-021-00164-4. PMID 34845569